CLINICAL TRIAL: NCT07035665
Title: A Single-Center, Randomized, Open-Label, Crossover Clinical Study to Evaluate the Effect of Food on the Pharmacokinetic Profiles of HRS-5965 Capsules in Healthy Subjects
Brief Title: A Clinical Study to Evaluate the Effect of Food on the Pharmacokinetic Profiles of HRS-5965 Capsules in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-108
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: IgA Nephropathy; Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Glomerulonephritis, IGA; Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-5965 Group A (Experimental)
  Interventions: Drug: HRS-5965 Capsules
- HRS-5965 Group B (Experimental)
  Interventions: Drug: HRS-5965 Capsules

INTERVENTIONS:
Drug: HRS-5965 Capsules — Oral doses of HRS-5965 capsules at fasted and fed conditions.

SUMMARY:
The study is being conducted to evaluate the effect of food on pharmacokinetics of HRS-5965 capsules after oral administration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form pre-trial.
2. Aged 18-45 years at signing the informed consent form.
3. Childbearing potential subjects: no pregnancy/sperm/egg donation plans; effective contraception.

Exclusion Criteria:

1. Recent infection (≤2 weeks): pathogen-positive test, systemic antibiotics, or fever > 38°C.
2. Major trauma/surgery (≤8 weeks) or planned surgery during the study.
3. Drug abuse history or positive urine drug screen.
4. Investigator-assessed suitability concerns: increased risk, compliance issues, or clinical ineligibility.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) of HRS-5965 | Day 1 to Day 13.
Area under the plasma concentration - time curve from time 0 to the last quantifiable timepoint (AUC0-t) | Day 1 to Day 13.

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) | Day 1 to Day 13.
Adverse events (AEs) | Day 1 to Day 20.

CONTACTS AND LOCATIONS:
Locations (1):
- ZhongShan Hospital FuDan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided